CLINICAL TRIAL: NCT04993508
Title: Randomized Prospective Multi Center Cohort Study for Primary Diagnosis of Clinically Significant Prostate Cancer With Combination of PSA/DRE and Multi Parametric Magnetic Resonance Imaging
Acronym: PRIMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital, Aachen (Other); University Hospital, Bonn (Other); University Hospital of Cologne (Other); University Hospital, Essen (Other); University Hospital Muenster (Other); German Cancer Research Center (Other); Marienhospital Herne (Other); Städtische Kliniken Mönchengladbach (Unknown); Evangelische Kliniken Essen-Mitte (Unknown); Klinikum Dortmund (Unknown); Stiftungsklinikum PROSELIS gGmbH Recklinghausen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-1389
Record Dates: First submitted 2021-06-08; First posted 2021-08-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate cancer diagnosis; multiparametric Magnetic Resonance Imaging (mpMRI); detection of clinically significant prostate cancer; avoidance of over diagnosis; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Men with PI-RADS 4/5 or PI-RADS 3 in conjunction with PSAD ≥ 0.15 that are randomized into arm A will undergo only targeted MRI/US fusion-guided biopsies. Men with PI-RADS 3 and PSAD > 0.15 with negative biopsy results will receive a follow-up MRI after 12 months. In case of upgrade to PI-RADS 4/5, men will be re-biopsied. Men with PI-RADS 4/5 without cancer diagnosis or with clinically insignificant cancer in the subsequent biopsy will be offered an additional MRI inbore biopsy. If MRI inbore biopsy is negative or with clinically insignificant cancer, men will be followed-up with MRI after 12 months. In the case of persistent PI-RADS 4/5, men will be re-biopsied.
  Interventions: Diagnostic Test: PSA test; Device: multiparametric prostate Magnetic Resonance Imaging (mpMRI); Procedure: targeted MRI/US fusion-guided biopsy; Procedure: MRI inbore biopsy
- Arm B (Active Comparator): Men with PI-RADS 4/5 or PI-RADS 3 in conjunction with PSAD ≥ 0.15 that are randomized into arm B will undergo targeted MRI/US fusion-guided biopsies and systematic biopsies (standard of care). Men with PI-RADS 3 and PSAD > 0.15 with negative biopsy results will receive a follow-up MRI after 12 months. In case of upgrade to PI-RADS 4/5, men will be re-biopsied. Men with PI-RADS 4/5 without cancer diagnosis or with clinically insignificant cancer in the subsequent biopsy will be offered an additional MRI inbore biopsy. If MRI inbore biopsy is negative or with clinically insignificant cancer, men will be followed-up with MRI after 12 months. In the case of persistent PI-RADS 4/5, men will be re-biopsied.
  Interventions: Diagnostic Test: PSA test; Device: multiparametric prostate Magnetic Resonance Imaging (mpMRI); Procedure: combined prostate biopsy (systematic biopsy plus targeted MRI/US fusion-guided biopsy); Procedure: MRI inbore biopsy

INTERVENTIONS:
Diagnostic Test: PSA test — testing for blood levels of PSA
Device: multiparametric prostate Magnetic Resonance Imaging (mpMRI) — mpMRI acquisition and reporting will be performed according to the current version of the Prostate Imaging-Reporting and Data System (PI-RADS). MpMRI will be performed at the different study centers on a 3 Tesla MR scanner using multi-phased array surface coil. MpMRI includes T1-weighted and T2-weighted imaging (T1WI, T2WI), diffusion-weighted imaging (DWI), and dynamic contrast-enhanced imaging (DCE-MRI). Hyoscine butyl bromide will be administered to optimize image quality. Prostate imaging quality will be assessed by the prostate imaging quality score (PI-QUAL). In case of contraindications to MRI contrast agents, DCE will be omitted. In case of contraindications to hyoscine butyl bromide, it will be omitted. Lesions with a PI-RADS score of ≥ 4 and 3 with PSAD > 0.15 will considered suspicious for csPCa.
Procedure: targeted MRI/US fusion-guided biopsy — Targeted MRI/US fusion-guided biopsy (TB) are performed using transrectal ultrasound (max. 4 cores from 3 targets). MRI/US fusion-guided biopsies can be performed transrectally or transperineally. Ultrasound-guided biopsies will be performed with a 3-D probe and with local or general anesthesia. Coverage with antibiotics has to be provided as per local standard of care for all biopsies.
  Arms: Arm A
Procedure: combined prostate biopsy (systematic biopsy plus targeted MRI/US fusion-guided biopsy) — The combined biopsy comprises systematic biopsy (SB) and targeted MRI/US fusion-guided biopsy (TB). They are performed using transrectal ultrasound (number of cores: SB 12 cores, TB max. 4 cores from 3 targets). MRI/US fusion-guided biopsies can be performed transrectally or transperineally. Ultrasound-guided biopsies will be performed with a 3-D probe and with local or general anesthesia. Coverage with antibiotics has to be provided as per local standard of care for all biopsies.
  Arms: Arm B
Procedure: MRI inbore biopsy — MRI inbore biopsies will be offered after negative initial MRI/US fusion-guided biopsy or diagnosis of only clinically insignificant PCa in initial biopsy in arms A or B. Before performing MRI inbore biopsy the PI-RADS scoring will be re-confirmed. The number of cores will be 2 per target. In case of inaccurate needle position additional cores are allowed to ensure correct targeting. Needle position will be verified in 2 planes. Coverage with antibiotics has to be provided as per local standard of care.

SUMMARY:
This randomized prospective multi center study is designed to confirm a new diagnostic pathway in primary diagnosis of clinically significant prostate cancer by combination of serum levels of prostate specific antigen (PSA), digitorectal examination (DRE), and multiparametric magnetic resonance imaging (mpMRI). Men at the age of 50 to 75 with an elevated PSA (>= 3 ng/ml) and /or suspicious DRE receive an upfront multi parametric MRI. Only men with MRI results suspicious of clinically significant prostate cancer will be biopsied. Those will be randomized into arm A and arm B. Arm A undergoes only targeted MRI/US fusion-guided biopsies (= TB with a maximum of 3 targets and 4 cores per target). Arm B receives systematic biopsies (= SB with 12 biopsy cores) and TB. Men with unsuspicious mpMRI will be receive follow-up according to current clinical standards. PRIMA will prospectively evaluate if stand-alone targeted MRI/US fusion-guided biopsy alone is sufficient to detect clinically significant prostate cancer (csPC with (ISUP grade group ≥ 2) and to avoid unnecessary detection of low-grade PC (ISUP 1) in biopsy-naïve men compared to a combined biopsy (systematic plus targeted) approach. The results of this study will directly influence clinical practice, will have a positive impact on patients' lives, and will lower the financial burden due to reduced overdiagnosis and over treatment.

DETAILED DESCRIPTION:
Men at the age of 50 to 75 years with an elevated PSA (≥ 3 ng/ml) and/or suspicious DRE receive a multiparametric MRI (mpMRI) and will be stratified based on MRI results. Only men with suspicious MRI, PI-RADS 4/5, and PI-RADS 3 in conjunction with high PSA density (PSAD > 0.15) are biopsied.

These will be randomized into arms A nd B. While patients in arm A undergo only targeted MRI/US fusion-guided biopsies (TB), patients in the "combined" arm B receive systematic biopsies (SB) and TB.

Statistical analysis for the detection rate of clinically significant and insignificant prostate cancers is composed of testing the non-inferiority and superiority of TB vs. TB+SB, respectively, using a global significance level of α = 0.05.

Interventions that are conducted within the PRIMA trial include PSA testing, digital rectal examination of the prostate (DRE), multiparametric prostate MRI, systematic and MRI/US fusion-guided biopsies as well as MRI inbore biopsies.

Arms A + B: Men with PI-RADS 4/5 and PI-RADS 3 in conjunction with PSAD > 0.15 will be randomized into arm A or arm B and biopsied as explained above. Men with PI-RADS 3 and PSAD > 0.15 with negative biopsy results will receive a follow-up MRI after 12 months. In case of upgrade to PI-RADS 4/5, men will be re-biopsied. Men with PI-RADS 4/5 without cancer diagnosis or with clinically insignificant cancer in the subsequent biopsy will be offered an additional MRI inbore biopsy. If MRI inbore biopsy is negative or with clinically insignificant cancer in men with PI-RADS 4/5, men will be followed-up with MRI after 12 months. In the case of persistent PI-RADS 4/5, men will be re-biopsied.

ELIGIBILITY:
Inclusion Criteria:

* Men aged from 50 to 75 years
* elevated PSA ≥ 3 ng/ml and/or cancer suspicious DRE

Exclusion Criteria:

* Men with known prostate cancer
* men with prior prostate biopsy
* men with non-MRI compatible devices
* men with acute prostatitis

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1908 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
detection rate of clinically significant and insignificant prostate cancers | 48 months
  The composite primary endpoint comprises non-inferiority in detecting clinically significant prostate cancer (ISUP grade group ≥ 2) and superiority in avoiding detection of clinically insignificant prostate cancer (ISUP grade group 1) of TB (arm A) compared to TB+SB (arm B)

SECONDARY OUTCOMES:
Pain score (Visual Analogue Scale [VAS]) | 48 months
  Patient Reported Outcomes (PROs) - diagnostic burden in arm A and B
Patient Reported Outcomes (PROs) - complications after biopsy | 30-day
  30-day complication-rate after biopsy in arm A and B
Patient Reported Outcomes (PROs) - quality of life according to EORTC-QLQ-C30 | 48 months
  quality of life according to EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life of Cancer Patientes; Scoring according to manual) in all different study arms
Patient Reported Outcomes (PROs) - quality of life according to EPIC-26 | 48 months
  quality of life according to EPIC-26 (Expanded prostate cancer index composite; Scoring according to manual) in all different study arms
number of biopsies avoided | 48 months
  Number of biopsies avoided with pre-biopsy mpMRI
detection rate of MRI inbore biopsy | 48 months
  Detection rate of MRI inbore biopsy after negative TB
detection rate of biparametric MRI | 48 months
  Detection rate of biparametric MRI (no perfusion imaging)
Number of up- and downgrading of PI-RADS score | 48 months
  Number of up- and downgradings of PI-RADS (Prostate Imaging - Reporting and Data System) score in follow-up mpMRIs
IPSS | 48 months
  International Prostate Symptom Score
IIEF-6 | 48 months
  International Index of Erectile Function

CONTACTS AND LOCATIONS:
Overall Officials: Rouvier Al-Monajjed, MD, Principal Investigator — Heinrich Heine University Düsseldorf / Urology; Lars Schimmöller, MD, Principal Investigator — Heinrich Heine University Düsseldorf / Radiology; Peter Albers, MD, Study Chair — Heinrich Heine University Düsseldorf / Urology; Gerald Antoch, MD, Study Chair — Heinrich Heine University Düsseldorf / Radiology; Matthias Boschheidgen, MD, Study Chair — Heinrich Heine University Düsseldorf / Radiology; Jan Philipp Radtke, MD, Study Chair — Heinrich Heine University Düsseldorf / Urology; Axel Benner, Study Chair — German Cancer Research Center / Biostatistics; Boris Hadaschik, MD, Study Chair — University Hospital Essen / Urology

IPD SHARING:
Plan to Share IPD: No